CLINICAL TRIAL: NCT06178757
Title: Comparison of Ultrasound-Guided Transversus Abdominis Plane Block (TAP) and External Oblique Plan Block (EOIB) for Postoperative Recovery and Pain Scores After Laparoscopic Cholecystectomy Surgery
Brief Title: TAP Block vs External Oblique Plane Block for Laparoscopic Cholecystectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 35
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cholecystitis; Cholecystitis, Acute; Cholecystitis, Chronic
Keywords: Laparoscopic Cholesistectomy; Postoperative pain management; External oblique intercostal block; Transversus abdominis plane block
MeSH Terms: conditions — Cholecystitis; Cholecystitis, Acute; Bronchiolitis Obliterans Syndrome | interventions — 1,3-bis(4-amidinophenoxy)-2-(4-amidinophenoxymethyl)ethylpropane

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for laparoscopic cholecystectomy surgery will be included in the study. Patients will be randomly divided into two groups (Group TAPB = TAP group, Group EOIB = EOB group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TAPB = Transversus abdominis plane block group (Active Comparator): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. 0,5 mg/kg meperidin will be performed for rescue analgesia
  Interventions: Drug: TAPB
- Group EOIB = External oblique intercostal plane block group (Active Comparator): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. 0,5 mg/kg meperidin will be performed for rescue analgesia
  Interventions: Drug: EOIB

INTERVENTIONS:
Drug: TAPB — As soon as the surgical procedure is completed, TAPB will be applied before extubation. After aseptic conditions are ensured, the high-frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The US probe will be placed at the level of the anterior axillary line between the 12th rib and the iliac crest, and the external oblique abdominal muscle, internal oblique abdominal muscle, and transverse abdominis muscle will be visualized. Then, using the in-plane technique, the needle will be advanced with the help of ultrasound until the needle tip reaches the space between the internal oblique and transversus abdominis muscles. After negative pressure aspiration, 5ml saline will be injected and the block location will be confirmed. Once the block location is confirmed, 20ml 0.25% bupivacaine (40ml total for each side) will be injected bilaterally.
  Arms: Group TAPB = Transversus abdominis plane block group
Drug: EOIB — As soon as the surgical procedure is completed, EOIB will be applied before extubation. After aseptic conditions are ensured, the high-frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath in the supine position, and an 80 mm block needle (Braun 360°) will be used. The US probe will be placed on the 6th rib in the mid-axillary line, at the line between the anterior superior iliac spine and the umbilicus. Using the In-Plane technique, 5 ml of saline will be injected between, the external oblique muscle and the rib, and the block location will be confirmed. After confirming the block location, 20 ml 0.25% bupivacaine will be applied to the plane between 6.,7., and 8. ribs and the muscles. The same procedure will be applied to the other side (a total of 40 ml 0.25% bupivacaine).
  Arms: Group EOIB = External oblique intercostal plane block group

SUMMARY:
Ultrasound (US) guidedTransversus Abdominis Plane Block (TAPB) is performed by injecting a local anesthetic into the plane between the internal oblique and transverse abdominis muscles and provides analgesia in the anterolateral walls of the abdomen after abdominal surgery. Ultrasound-guided TAPB has been commonly used for many years.

US-guided External oblique intercostal block (EOIB) is a novel block performed by injection of local anesthetic between the external and internal oblique muscles at the level of 6th-8th ribs. This block provides abdominal analgesia between T6 and T10 levels. There are studies in the literature showing that it provides effective analgesia. However, there is no study comparing TAPB and EOIB yet.

In this study, we aim to compare the effectiveness of US-guided TAPB and EOIB for postoperative analgesia management after laparoscopic cholecystectomy surgery. Our primary aim is to compare patient recovery scores (QoR15 Turkish version), our secondary aim is to compare postoperative pain scores (24-hour NRS), postoperative rescue analgesic use (opioid/meperidine), and opioid-related side effects (allergic reaction, nausea, vomiting).

DETAILED DESCRIPTION:
Cholecystectomy is the most common abdominal surgery performed in developed countries and is usually performed laparoscopically. The etiology of pain after laparoscopic cholecystectomy is multifactorial and is generally considered visceral pain. Diaphragmatic nerve irritation due to CO2 insufflation into the peritoneal cavity, abdominal distension, tissue damage, damage due to dissection of the gallbladder, sociocultural situation, and individual factors play a role in the occurrence of this pain..

Postoperative pain is an acute pain that is accompanied by inflammation caused by surgical stress and decreases over time with tissue healing. Pain in the postoperative period in patients undergoing laparoscopic cholecystectomy surgery is a serious problem that reduces patient comfort and delays the patient's return to work after surgery (4). Successful postoperative analgesia management prevents many of the complications such as respiratory problems and delayed mobilization (5).

Transverse Abdominis Plane Block (TAPB), performed under ultrasound (US) guidance, is a block that is performed by injecting a local anesthetic into the plane between the internal oblique and transverse abdominis muscles and provides analgesia in the anterolateral walls of the abdomen after surgery. Ultrasound-guided TAPB is commonly used.

TAPB provides analgesia in the abdominal region in T6-L1 dermatomes. Sonoanatomy is easy to visualize on US and the spread of local anesthetic can be seen. Analgesia occurs in several dermatomes with the cephalo-caudal spread of the local anesthetic solution. Studies are proving that TAP block is effective in some abdominal surgeries such as hysterectomy, cesarean section, cholecystectomy, inguinal hernia and prostatectomy. Sensory block areas formed by TAPB are highly variable and may result in insufficient blocks.

External oblique block (EOIB) performed under US guidance is a block performed by injection of local anesthetic between the external and internal oblique muscles. This block provides abdominal analgesia covering the T6-T10 dermatomes. There are studies in the literature proving that it provides effective analgesia (12-14). However, no study comparing TAPB and EOIP has been published yet.

In this study, we aim to compare the effectiveness of US-guided TAPB and EOIB for postoperative analgesia management after laparoscopic cholecystectomy surgery. Our primary aim is to compare patient recovery scores (QoR15 Turkish version), our secondary aim is to compare postoperative pain scores (24-hour NRS), postoperative rescue analgesic use (opioid/meperidine), and opioid-related side effects (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for laparoscopic cholecystectomy surgery under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* anticoagulant treatment
* local anesthetics and opioid allergy
* Infection at the site of the block
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Global recovery scoring system (patient satisfaction scale) | Change from baseline score at postoperative 24 hour
  We will use the Turkish version of Quality of Recovery / QoR-15 questionairre

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | Postoperative 24 hours period
  Change from Baseline Pain Scores at Postoperative 24 hours.
The use of rescue analgesia | Postoperative 24 hours period
  Meperidine using (Number of Participants and Concentration of Meperidine)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Elsharkawy H, Kolli S, Soliman LM, Seif J, Drake RL, Mariano ER, El-Boghdadly K. The External Oblique Intercostal Block: Anatomic Evaluation and Case Series. Pain Med. 2021 Nov 26;22(11):2436-2442. doi: 10.1093/pm/pnab296. PMID 34626112
- [Background] Hamilton DL, Manickam BP, Wilson MAJ, Abdel Meguid E. External oblique fascial plane block. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100256. doi: 10.1136/rapm-2018-100256. Online ahead of print. No abstract available. PMID 30635518
- [Background] Tulgar S, Ahiskalioglu A, Selvi O, Thomas DT, Ozer Z. Similarities between external oblique fascial plane block and blockage of thoracoabdominal nerves through perichondral approach (TAPA). J Clin Anesth. 2019 Nov;57:91-92. doi: 10.1016/j.jclinane.2019.03.027. Epub 2019 Mar 29. No abstract available. PMID 30933854